CLINICAL TRIAL: NCT05394233
Title: Efficacy and Safety of Tislelizumab Combined With Bevacizumab and Platinum Plus Pemetrexed for Untreated EGFR+ and High PD-L1 Expression Non-squamous NSCLC :a Phase II, Single-center, Single Arm Study
Brief Title: Tislelizumab +Bevacizumab+pc for Untreated EGFR+ and High PD-L1 Non-squamous NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Juan LI, MD, Director of standard treatment department of medical oncology, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAT1706-LJ2022
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Non-squamous Non-small Cell Lung Cancer; EGFR Gene Mutation
MeSH Terms: interventions — Bevacizumab; Platinum; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tislelizumab combined with bevacizumab and platinum plus pemetrexed (Experimental): Drug:
  Induction Phase:
  Bevacizumab: 7.5 mg/kg administered as an IV infusion on Day 1 of each 3-week cycle for 4 cycles Cisplatin 75 mg/m2 will be administered as an intravenous infusion over 2 hours every 3 weeks for 4 cycles.
  Pemetrexed, 500 mg/m2, intravenously, every 3 weeks for 4 cycles
  Maintenance phase:
  Tislelizumab, 200 mg IV every 3 weeks;until disease progression or intolerance Bevacizumab: 7.5 mg/kg administered as an intravenous infusion on Day 1 of each 3-week cycle;until disease progression or intolerance
  Interventions: Drug: Tislelizumab Combined With Bevacizumab and Platinum Plus Pemetrexed

INTERVENTIONS:
Drug: Tislelizumab Combined With Bevacizumab and Platinum Plus Pemetrexed — Bevacizumab: 7.5 mg/kg administered as an intravenous infusion on Day 1 of each 3-week cycle Cisplatin 75 mg/m2 will be administered as an intravenous infusion over 2 hours, every 3 weeks, Pemetrexed, 500 mg/m2, intravenously every 3 weeks, Tislelizumab, 200 mg IV every 3 weeks

SUMMARY:
A study to evaluate the efficacy and safety of tislelizumab combined with bevacizumab and platinum-based pemetrexed in the treatment of naïve patients with advanced non-squamous non-small cell lung cancer with sensitive EGFR mutations and high PD-L1 expression Prospective, open-label, single-arm phase II clinical study

DETAILED DESCRIPTION:
A study to evaluate the efficacy and safety of tislelizumab combined with bevacizumab and platinum-based pemetrexed in the treatment of naïve patients with advanced non-squamous non-small cell lung cancer with sensitive EGFR mutations and high PD-L1 expression Prospective, open-label, single-arm phase II clinical study;

Research purposes:

Main purpose: To evaluate the median progression-free rate of tislelizumab combined with bevacizumab and platinum pemetrexed in treatment-naïve advanced non-small cell lung cancer patients with sensitive EGFR mutations and high PD-L1 expression Survival (middle progression free survival, mPFS)

Secondary purpose:

* Evaluation of objective response rate (ORR) according to RECIST version 1.1;
* Evaluation of disease control rate (DCR) according to RECIST version 1.1;
* Assess overall survival (OS);
* Assess Duration of Response (DOR);
* Evaluate the safety of the treatment using NCI-CTCAE v5;

Exploratory Purpose:

• Assess potential predictive biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 and ≤ 75 years of age. Signed the informed consent form prior to patient entry
2. Histologically or pathologically confirmed non-squamous non-small cell lung cancer(NSCLC) with stage IV /III
3. Patients with EGFR sensitive mutations: 19del and L858R who have not been treated with TKI for the first time, the patients need to provide the test results of the certified detection platform, and the PD-L1 expression based on tissue specimen detection is greater than 50% (PD-L1 detection clone number: SP263).
4. A World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) Performance Status Score (PS) of 0 or 1 at the time of recruitment.
5. Adequate organ and bone marrow function, defined as:

   * Hemoglobin≥9.0 g/dL
   * Absolute neutrophil count ≥1.5 × 109/L
   * Platelet count ≥100 × 109/L
   * Serum bilirubin ≤ 1.5 × upper limit of normal range (ULN). This does not apply to patients diagnosed with Gilbert's syndrome (persistent or recurrent hyperbilirubinemia [primarily unconjugated bilirubin] without evidence of hemolysis or liver pathology), which may be allowed after consultation with a physician patients participating in the study.
   * ALT and AST ≤2.5 × ULN
   * Measured creatinine clearance (CL) >40 mL/min or Cockcroft-Gault calculated CL >40 mL/min (using actual body weight) Men: Creatinine clearance (mLmin⁄) = body weight (kg) x (140-age) 72 x serum creatinine (mg/dL) Female: creatinine clearance (mLmin⁄) = body weight (kg) x (140-age) 72 x serum creatinine (mg/dL) x 0.85
6. The expected survival time of patients is ≥3 months
7. Weight > 30 kg
8. Have the ability to sign the informed consent form and comply with the requirements and restrictions listed in the informed consent form (ICF) and this protocol.

Exclusion Criteria:

1. Patients with grade ≥2 non-infectious pneumonia.
2. History of allogeneic organ transplantation, except corneal transplantation.
3. Active or previously documented autoimmune or inflammatory diseases (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [except diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatous vasculitis, Graves disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). Exceptions to this standard include:

   * Vitiligo or alopecia patients
   * Patients with hypothyroidism who are stable on hormone replacement therapy (eg, after Hashimoto's syndrome)
   * Any chronic skin disease that does not require systemic treatment
   * Patients without active disease within the past 5 years may be included in the study, but only after consultation with the study physician
   * Patients with celiac disease that can be controlled with diet alone
4. Uncontrolled concurrent diseases, including but not limited to: persistent or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled arrhythmia, active ILD , Severe chronic gastrointestinal disease with diarrhea, or a psychiatric/social condition that may limit compliance with study requirements, cause a significantly increased risk of AEs, or interfere with the subject's ability to provide written informed consent.
5. History of another primary malignant tumor, except for the following cases;

   * Malignant tumors with low potential risk of recurrence and no known active disease ≥5 years prior to first dose treated with curative intent
   * Adequately treated non-melanoma skin cancer with no evidence of disease or lentigo maligna
   * Adequately treated cervical carcinoma in situ without evidence of disease
6. History of active primary immunodeficiency
7. Active infection, including tuberculosis (clinical assessment, including clinical history, physical examination, radiographic findings, and tuberculosis testing consistent with local clinical practice).
8. Known history of human immunodeficiency virus (HIV) infection; known active syphilis infection.
9. Untreated active hepatitis B

   Hepatitis B patients who meet the following criteria are eligible for inclusion:

   - Hepatitis B virus (HBV) load was below the lower limit of detection in our hospital before the first dose, and received anti-HBV therapy throughout the study period to avoid viral reactivation.
10. Subjects with active hepatitis C (HCV) infection, HCV antibody positive patients only meet the study inclusion criteria when the polymerase chain reaction of HCV RNA is negative.
11. Active brain metastases or spinal cord compression. Prior to study entry, all patients underwent MRI (preferred) or CT examination, preferably brain examination with intravenous contrast.
12. Known allergy or hypersensitivity reaction to any study drug or any study drug excipients
13. Previous exposure to immune-mediated therapy, including but not limited to: anti-PD-1, anti-PD-L1 and anti-programmed death ligand 2 (anti-PD-L2) antibodies, except for therapeutic anti-tumor vaccines .
14. Live attenuated vaccine should be vaccinated within 30 days before the first dose, and live vaccine should not be vaccinated within 30 days after the last dose.
15. Major surgery (as defined by the investigator) within 42 days prior to the first dose.
16. Within 14 days before administration, immunosuppressive drugs are being used or have been used in the past. Exceptions to this standard include:

    * Intranasal, inhaled, topical steroids, or topical steroid injections (eg, intra-articular injections)
    * Systemic corticosteroid therapy not exceeding 10 mg/day of prednisone or its physiologic equivalent
    * Steroids administered as prophylactic for hypersensitivity reactions (eg, prophylactic administration of CT scan)
17. Pregnant or lactating female patients and fertile male or female patients are unwilling to take effective contraceptive measures from screening to 6 months after the last dose.
18. Other researchers think that it is not suitable for inclusion.
19. Mixed cell lung cancer: non-small cell and small cell mixed lung cancer and mixed adenosquamous lung cancer dominated by squamous cell carcinoma.
20. Non-squamous non-small cell lung cancer with hemoptysis (>50 ml/day); clinically significant hemoptysis or bleeding symptoms occurred within 3 months before enrollment.
21. Patients with brain metastases whose symptoms are not controlled after treatment.
22. Imaging (CT/MRI) shows that the tumor lesion is less than 5 mm away from the large blood vessels, there is a central tumor that invades the local large blood vessels and is less than 2 cm away from the bronchial tree; or there is an obvious lung cavity or necrotic tumor.
23. Arterial/venous thrombotic events that occurred within 12 months before enrollment
24. Patients with any severe and/or uncontrolled disease (hypertension, liver cirrhosis, heart failure, etc.)
25. Major surgical operation or severe traumatic injury, fracture or ulcer occurred within 4 weeks before enrollment
26. Severe weight loss (greater than 10%)
27. Abnormal coagulation function, with bleeding tendency or receiving thrombolytic or anticoagulation therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
middle progression free survival | Estimated about 6 months
  To evaluate the median progression-free survival (middle) of tislelizumab combined with bevacizumab and platinum-based pemetrexed in treatment-naïve advanced non-small cell lung cancer patients with sensitive EGFR mutations and high PD-L1 expression. progression free survival (mPFS)

CONTACTS AND LOCATIONS:
Overall Officials: juan li, Study Director — Sichuan Cancer Hospital Chengdu, Sichuan China
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No